CLINICAL TRIAL: NCT07217327
Title: DistaSense: Two-Center Prospective, Non-Significant Risk (NSR) Study to Evaluate Heart Rate and Respiratory Rate Performance for Life Detection Technologies
Brief Title: The DistaSense VITALS Study
Acronym: VITALS
Status: Recruiting | Type: Observational
Sponsor: Life Detection Technologies (Industry)
Collaborators: Nilo Medical Consulting Group (Unknown)
Responsible Party: Sponsor
Other Study IDs: TP-25-002
Record Dates: First submitted 2025-07-30; First posted 2025-10-15 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-09

CONDITIONS: Detection of Heart Rate and Respiratory Rate
MeSH Terms: interventions — Polysomnography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: DistaSense and Polysomnography — All subjects will be evaluated by DistaSense and reference device for respiratory rate and heart rate.

SUMMARY:
A prospective, non-significant risk study designed to validate the performance of the DistaSense Contactless Sensor and algorithm for detecting heart rate and respiratory rate, compared to gold standard reference technology.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 22 years
2. Fluent in English
3. Willing and cognitively able to provide informed consent
4. BMI < 36
5. Expected by the investigator to achieve sufficient sleep duration for a minimum of 4 hours of meaningful data (e.g., absence of significant insomnia)
6. Able to complete the scripted portion of the evaluation

Exclusion Criteria:

1. Pregnant
2. Sufficiently broken, damaged or irritated skin or rashes near the sensor application sites such that investigator believes should be precluded from enrollment
3. Subjects with electronic implants of any kind (e.g. pacemaker)
4. Subjects that are Life Detection Technology employees or shareholders, or family of a Life Detection Technology employee or shareholder

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteers will be recruited via research subject databases from each site.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-08-13 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Accuracy and bias between the DistaSense measurements of heart rate and respiratory rate and the reference measurements | Day 1

SECONDARY OUTCOMES:
Mean absolute relative difference for each of HR and RR between the DistaSense and the reference | Day 1
Deming regression for each of the HR and RR data | Day 1

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Clayton Sleep Institute, St Louis, Missouri
  - CTI Clinical Research Center, Cincinnati, Ohio